CLINICAL TRIAL: NCT06264037
Title: "The Experiences of Care Lived by People Admitted to Neurorehabilitation: a Qualitative Exploratory Study With a Phenomenological Approach
Brief Title: The Experience in Neurorehabilitation Setting: a Qualitative Study
Acronym: NURSEXPERIENCE
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.03; Studio 1574 /IRCCS San Camillo (Other: CESC di Venezia e IRCSS San Camillo)
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Rehabilitation; Neurologic Disorder; Stroke; Parkinson Disease; Multiple Sclerosis; Neurosurgery
MeSH Terms: conditions — Nervous System Diseases; Stroke; Parkinson Disease; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with stroke: Patients with stroke during the hospital neurorehabilitation
  Interventions: Other: semi structured interview
- People with Parkinson's disease: patients with Parkinson's disease the hospital neurorehabilitation
  Interventions: Other: semi structured interview
- Patients with multiple sclerosis: Patients with multiple sclerosis during the hospital neurorehabilitation
  Interventions: Other: semi structured interview
- Patients post operative oncological neuro surgery: Patients after oncological neurosurgical operation during the hospital neurorehabilitation
  Interventions: Other: semi structured interview

INTERVENTIONS:
Other: semi structured interview — semistructured interview on patient's experience of hospitalization.

SUMMARY:
In this exploratory qualitative study with a hermeneutic phenomenological approach, we will describe and understand the experience of treatment and hospitalization in hospitalized people suffering from stroke, multiple sclerosis, Parkinson's disease and patients post-neurosurgery for oncological causes. Patients will be interviewed in a semi-structured manner and sampling will take place for each of the pathology groups according to the saturation method.

DETAILED DESCRIPTION:
This is an exploratory qualitative study with a hermeneutic phenomenological approach on a cohort of patients hospitalized at San Camillo IRCCS.

Description of the study Type of patients: Patients in neurorehabilitation with stroke, Multiple Sclerosis, Parkinson's, post surgery in neurosurgery for oncological pathology. In fact, the recent systematic review on the topic of perception of well-being in elderly people with stroke admitted to neurorehabilitation by Lafiatoglu et al. (2022) highlights 5 themes in the literature that influence the perception of well-being in patients: rehabilitation processes; identity and self-perception problems; institutional factors; experience of caring and participation in other creative activities during hospitalization.

From another perspective, not referring to well-being, but to the hospitalization experience itself, the systematic review by Luker et al. (2015) examining 31 studies highlighted how all reported negative rehabilitation experiences, including helplessness, boredom and frustration, lack of control, lack of understanding and lack of effective communication. Rosewilliam et al. (2011) also point to negative experiences and various barriers that hinder the application of a patient-centered goal-setting model in stroke rehabilitation practice.

Finally, the review by Neils-Strunjas et al. (2017) explored the construct of resilience in the rehabilitation of adults with ABI concluding that resilience plays a vital role in the recovery and rehabilitation process by amplifying individuals' emotional adjustment and adjustment after ABI.

There appears to be less literature referring to patients with multiple sclerosis, although a trend has recently developed in Germany that welcomes the perspectives of patients in rehabilitation. The considerations of Gaidar et al appear important to us. (2022) and Geisler et al. (2020) who instead note the lack and consequently the need for patients with MS to be involved in decision making processes regarding their own care and rehabilitation as a major theme in the hospitalization experience, while other aspects present in patients with stroke , they don't seem to emerge.

There is a fair amount of literature dedicated to the life experiences of people suffering from Parkinson's disease (Soundy et al. 2014), however qualitative studies dedicated to the experiences of hospitalization in a rehabilitation context are very limited.

Even less described, again in the hospital rehabilitation setting, are the experiences of patients who have rehabilitation after neurosurgery (Loomis & Wakasa, 2020); focusing these either on the oncological aspects of experience or on the surgical and intensive care ones (Greenberg et al. 2006).

But the peculiarities of the life experience of this type of patients during hospital motor rehabilitation, often still bedridden, often still waiting for further oncological therapies, are not yet described.

Phenomenology refers to both a philosophical current and a research approach, it was founded by Husserl and subsequently developed by Heidegger. It aims to understand people's lived experience.

In our study it was decided to adopt a hermeneutic-interpretive approach because the researcher's posture during interviews based on epochè is difficult to maintain in a hospital context when the researchers still belong to the hospital staff itself.

Concretely, a typical qualitative and narrative research tool will be used [Charon, 2001; Winding & Whiteford, 2005; Pringle et al, 2011; Ambrosi & Canzan, 2013; Fleming et al, 2013]: specifically semi-structured interviews.

This choice will allow us to get as close as possible to understanding the meaning of the experience lived by the patients involved.

In fact, as is known, the object of the phenomenological gaze is not the experience in itself but the experience lived by a subject in a precise moment of his life and the personal meaning that it comes to take on for him and for his history. of life.

Razionale In neurorehabilitation, the literature agrees in giving great value to the hospitalization environment, as well as to the activities and the relationship, not necessarily focused on therapy, with the staff. This literature is particularly developed, mainly with qualitative studies, with patients suffering from ABI, Acquired Brain Injuries, in fact mainly stroke.

Objective:

The objective of this study is to describe and understand the experience of treatment and hospitalization in people admitted to neurorehabilitation suffering from stroke, multiple sclerosis, Parkinson's disease and patients post-neurosurgery for oncological causes.

Methods:

Patients admitted to neurorehabilitation who belong to the following pathologies will be selected according to sampling for saturation: stroke, multiple sclerosis, Parkinson's disease and post-neurosurgery for oncological causes. The patient who meets the inclusion and exclusion criteria, after 21 days of hospitalization which must have elapsed without transfers or acute phases even if treated within the IRCCS San Camillo, will be contacted by a researcher of the research project who will illustrate and will explain the research project in a comprehensive and comprehensible manner in order to obtain valid consent.

Once consent has been obtained, the best time to carry out the interview will be agreed with the patient, which will be semi-structured in nature and based on a grid of questions aimed at exploring the patient's hospitalization experience and perception of care.

A duration of approximately 45 minutes per interview is assumed. The interviews will be carried out by specially trained researchers. To test the semi-structured interview grid, four to five pilot interviews will be carried out which will not then be part of the sample to be analyzed with content analysis.

Given the scarcity of literature on the topic, with the exception of that relating to patients hospitalized in neurorehabilitation with stroke, the pilot interview phase will also serve to refine the interview grid.

The analysis of the interviews will take place with the content analysis software Atlas ti© (22 or 23).The variables referring to socio-demographic and clinical data and those referring to the Barthel and FIMM scales will be treated using descriptive statistics. Specifically, the normally distributed variables will be presented using the mean and standard deviation, the variables with asymmetric distribution will be presented using the median and interquartile range, while the categorical variables by means of absolute values and frequencies.

The analysis of the narrative material of the interviews will take place according to the following phases.

1. Pre-analysis phase:

   All the collected text will be transcribed verbatim into a word file, then read repeatedly by the researchers to familiarize themselves with the material (holistic reading) and arrive at an overall vision; then introduced in "Atlas ti" (22 or 23) (Scientific Software Development GmbH, Berlin, Germany), a computer program developed to aid the coding process in qualitative research that belongs to the CAQDAS category.
2. Material exploration phase:

   In this phase all the material is processed by the Atlas ti software which creates hermeneutic units and quotations which will serve as a basis in the analysis of the codes and families that arise from the processing of the Hermeneutic Units. . In this phase the coding work will be carried out by two researchers who will independently proceed with the analysis according to a method consistent with the Gadamerian "art of texting".
3. Interpretation phase In this phase the final coding structure, and the raw data it contains, is processed in order to restore meaning and validity, allowing the researcher to organize the results in tables, diagrams, figures, or by creating a network that shows the deducible relationships between the codes inside families It is not possible to indicate a priori a sample size given the choice of saturation sampling. 10 per cohort are assumed.

As Expected Results are expected Identification of the most relevant themes and aspects to consider during hospitalization to carry out neurological rehabilitation.

Description of experiences lived by people hospitalized in neurological rehabilitation Identification of factors that can contribute to making hospitalization pleasant.

Formulation of new hypotheses to explore the relationship between hospitalization experience and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:● Patients hospitalized at the IRCCS San Camillo.

* patients in Stroke, Multiple Sclerosis, Parkinson's Disease and post-operative patients in Neurosurgery for oncological pathology
* Patients who have given valid consent.
* Patients able to understand, read and speak Italian.
* Aphasic patients without comprehension deficits and able to communicate effectively with augmented communication media.
* hospitalized for at least 21 days and not close to discharge, or that this occurs at least after 21 days.

Exclusion Criteria:● Patients unable to give valid consent.

* Minor patients or patients over 85 years of age.
* Patients with cognitive deficits such that they cannot effectively support the interview.
* Patients with psychiatric pathology
* Patients unable to understand, read and speak Italian.
* Patients with pathologies for which they are not undergoing neurorehabilitation treatment.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Stroke, Multiple Sclerosis, Parkinson's Disease and post-operative Neurosurgery patients admitted to the IRCCS San Camillo will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-12-08 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
narrative contents | 30- 40 minutes of interview
  the personal experience of hospital stay in neurorehabilitaion setting

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Camuccio, doctor, Principal Investigator — IRCCS San Camillo
Locations (3):
- Italy (3):
  - Alberto Camuccio, Venezia
  - IRCCS San Camillo Department of Neurorehabilitation, Venezia, Venezia
  - IRCCS San Camillo Venezia, Venezia

REFERENCES:
- [Result] Batbaatar E, Dorjdagva J, Luvsannyam A, Savino MM, Amenta P. Determinants of patient satisfaction: a systematic review. Perspect Public Health. 2017 Mar;137(2):89-101. doi: 10.1177/1757913916634136. Epub 2016 Jul 20. PMID 27004489
- [Result] Canzan F, Saiani L, Mortari L, Ambrosi E. [When patients talk about healing: a phenomenological qualitative study]. Assist Inferm Ric. 2013 Oct-Dec;32(4):205-12. doi: 10.1702/1381.15358. Italian. PMID 24441465
- [Result] Chen Y, Zhou W, Hou L, Zhang X, Wang Q, Gu J, Zhang R, Yang H. The subjective experience of family caregivers of people living with Parkinson's disease: a meta-ethnography of qualitative literature. Aging Clin Exp Res. 2022 May;34(5):959-970. doi: 10.1007/s40520-021-01995-9. Epub 2021 Oct 14. PMID 34648175
- [Result] Fidder H, Jaski JJ, Elbertse E, van Loon AM, Monnier AA, de Boer ME, de Groot AJ. Parkinson rehabilitation in nursing homes: a qualitative exploration of the experiences of patients and caregivers. Eur Geriatr Med. 2022 Oct;13(5):1197-1210. doi: 10.1007/s41999-022-00647-z. Epub 2022 May 11. PMID 35543902
- [Result] Fleming V, Gaidys U, Robb Y. Hermeneutic research in nursing: developing a Gadamerian-based research method. Nurs Inq. 2003 Jun;10(2):113-20. doi: 10.1046/j.1440-1800.2003.00163.x. PMID 12755860
- [Result] Ghaidar D, Sippel A, Riemann-Lorenz K, Kofahl C, Morrison R, Kleiter I, Schmidt S, Dettmers C, Schulz H, Heesen C. Experiences of persons with multiple sclerosis with rehabilitation-a qualitative interview study. BMC Health Serv Res. 2022 Jun 11;22(1):770. doi: 10.1186/s12913-022-08150-8. PMID 35690766
- [Result] Giesler JM, Klindtworth K, Nebe A, Glattacker M. [Medical Rehabilitation in MS: Barriers to and Facilitators of its Utilization from the Patients' Perspective]. Rehabilitation (Stuttg). 2020 Apr;59(2):112-119. doi: 10.1055/a-0965-0977. Epub 2019 Aug 13. German. PMID 31408893
- [Result] Greenberg E, Treger I, Ring H. Rehabilitation outcomes in patients with brain tumors and acute stroke: comparative study of inpatient rehabilitation. Am J Phys Med Rehabil. 2006 Jul;85(7):568-73. doi: 10.1097/01.phm.0000223218.38152.53. PMID 16788387
- [Result] Gualandi R, Masella C, Viglione D, Tartaglini D. Exploring the hospital patient journey: What does the patient experience? PLoS One. 2019 Dec 5;14(12):e0224899. doi: 10.1371/journal.pone.0224899. eCollection 2019. PMID 31805061
- [Result] Guest G, Namey E, Chen M. A simple method to assess and report thematic saturation in qualitative research. PLoS One. 2020 May 5;15(5):e0232076. doi: 10.1371/journal.pone.0232076. eCollection 2020. PMID 32369511
- [Result] Hennink M, Kaiser BN. Sample sizes for saturation in qualitative research: A systematic review of empirical tests. Soc Sci Med. 2022 Jan;292:114523. doi: 10.1016/j.socscimed.2021.114523. Epub 2021 Nov 2. PMID 34785096
- [Result] Loft MI, Martinsen B, Esbensen BA, Mathiesen LL, Iversen HK, Poulsen I. Call for human contact and support: an interview study exploring patients' experiences with inpatient stroke rehabilitation and their perception of nurses' and nurse assistants' roles and functions. Disabil Rehabil. 2019 Feb;41(4):396-404. doi: 10.1080/09638288.2017.1393698. Epub 2017 Oct 24. PMID 29065725
- [Result] Loomis E, Wakasa M. Rehabilitation from meningioma. Handb Clin Neurol. 2020;170:323-331. doi: 10.1016/B978-0-12-822198-3.00051-3. PMID 32586505
- [Result] Luker J, Lynch E, Bernhardsson S, Bennett L, Bernhardt J. Stroke Survivors' Experiences of Physical Rehabilitation: A Systematic Review of Qualitative Studies. Arch Phys Med Rehabil. 2015 Sep;96(9):1698-708.e10. doi: 10.1016/j.apmr.2015.03.017. Epub 2015 Apr 3. PMID 25847387
- [Result] Mangset M, Tor Erling Dahl, Forde R, Wyller TB. 'We're just sick people, nothing else': ... factors contributing to elderly stroke patients' satisfaction with rehabilitation. Clin Rehabil. 2008 Sep;22(9):825-35. doi: 10.1177/0269215508091872. PMID 18728136
- [Result] Moser A, Korstjens I. Series: Practical guidance to qualitative research. Part 3: Sampling, data collection and analysis. Eur J Gen Pract. 2018 Dec;24(1):9-18. doi: 10.1080/13814788.2017.1375091. Epub 2017 Dec 4. PMID 29199486
- [Result] Olofsson A, Andersson SO, Carlberg B. 'If only I manage to get home I'll get better'--interviews with stroke patients after emergency stay in hospital on their experiences and needs. Clin Rehabil. 2005 Jun;19(4):433-40. doi: 10.1191/0269215505cr788oa. PMID 15929513
- [Result] Panday J, Velikonja D, Moll SE, Harris JE. Experiences of inpatient rehabilitation from the perspective of persons with acquired brain injury. Disabil Rehabil. 2022 Sep;44(19):5539-5548. doi: 10.1080/09638288.2021.1938706. Epub 2021 Jun 24. PMID 34166176
- [Result] Sadrameli SS, Chan TM, Vaziri S, Murad GJA, Hooten KG. Patient-Reported Outcomes: Quality of Care on a Neurosurgical Ward. Qual Manag Health Care. 2021 Jul-Sep 01;30(3):194-199. doi: 10.1097/QMH.0000000000000284. PMID 33591084
- [Result] Soratto J, Pires DEP, Friese S. Thematic content analysis using ATLAS.ti software: Potentialities for researchs in health. Rev Bras Enferm. 2020 Apr 22;73(3):e20190250. doi: 10.1590/0034-7167-2019-0250. eCollection 2020. PMID 32321144
- [Result] Soundy A, Stubbs B, Roskell C. The experience of Parkinson's disease: a systematic review and meta-ethnography. ScientificWorldJournal. 2014;2014:613592. doi: 10.1155/2014/613592. Epub 2014 Nov 30. PMID 25525623
- [Result] Sundler AJ, Lindberg E, Nilsson C, Palmer L. Qualitative thematic analysis based on descriptive phenomenology. Nurs Open. 2019 Apr 7;6(3):733-739. doi: 10.1002/nop2.275. eCollection 2019 Jul. PMID 31367394
- [Result] Tholin H, Forsberg A. Satisfaction with care and rehabilitation among people with stroke, from hospital to community care. Scand J Caring Sci. 2014 Dec;28(4):822-9. doi: 10.1111/scs.12116. Epub 2014 Feb 5. PMID 24495250
- [Result] Tran VT, Porcher R, Tran VC, Ravaud P. Predicting data saturation in qualitative surveys with mathematical models from ecological research. J Clin Epidemiol. 2017 Feb;82:71-78.e2. doi: 10.1016/j.jclinepi.2016.10.001. Epub 2016 Oct 24. PMID 27789316
- [Result] Witzig-Brandli V, Lange C, Gschwend S, Kohler M. "I would stress less if I knew that the nurse is taking care of it": Multiple Sclerosis inpatients' and health care professionals' views of their nursing-experience and nursing consultation in rehabilitation-a qualitative study. BMC Nurs. 2022 Aug 23;21(1):232. doi: 10.1186/s12912-022-01013-x. PMID 35999594